CLINICAL TRIAL: NCT02686437
Title: Tension of THERABAND® Kinesiology Tape on Shoulder Pain
Acronym: ShoulderTBKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSR06
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Results first posted 2017-10-10 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-12

CONDITIONS: Shoulder Pain
Keywords: shoulder dysfunction; kinesiology tape; rehabilitation
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increasing Tension (Experimental): The kinesiology tape will be applied to the shoulder complex to influence proper activation of the rotator cuff muscles, specifically the supraspinatus and infraspinatus. The clinician applied the tape in an "I" strip from the vertebral border of the scapula to the lesser tubercle of the humerus. Over the course of the 4 weeks of care, the tension of the Intervention Group's tape will systemically increase based on the following timelines:
  Week 1: 0% tension Week 2: 25% tension Week 3: 50% tension Week 4: 75% tension
  Interventions: Other: TheraBand Kinesiology Tape
- Control Tension (Sham Comparator): The kinesiology tape will be applied to the shoulder complex to influence proper activation of the rotator cuff muscles, specifically the supraspinatus and infraspinatus. The clinician applied the tape in an "I" strip from the vertebral border of the scapula to the greater tuberosity of the humerus. Over the course of the 4 weeks of care, the tension of the Control Group's tape will remain at 0% tension
  Interventions: Other: TheraBand Kinesiology Tape

INTERVENTIONS:
Other: TheraBand Kinesiology Tape — Kinesiology taping technique is designed to target muscles and lymphatic system. Limited research is available for specific conditions, including low back pain, but it is theorized to correct muscle function by inhibiting or facilitating the muscle, improve blood flow, reduce pain, and improve joint alignment.

SUMMARY:
The purpose of this study is to determine the effectiveness of standard tension of Thera-Band® Kinesiological Tape (TB-KT) application versus varied tension on shoulder pain, disability, and recovery speed during an in-office rehabilitative program. A convenience sample size of 38 new patients with current shoulder pain will be recruited for this study. The outcome measures will include the Numeric Pain Rating Scale (NPRS) and the Penn Shoulder Score (PENN). After completing the initial paperwork, patients will be randomized into two groups, control (0% tension) and intervention(increasing tension). At the beginning of each week the tape will be reapplied, and pain rating will be recorded. At the conclusion of 4 weeks patients will complete the PENN.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of standard tension of Thera-Band® Kinesiological Tape (TB-KT) application versus varied tension on shoulder pain, disability, and recovery speed during an in-office rehabilitative program. A convenience sample size of 38 new patients with current shoulder pain will be recruited for this study. Patients must be tested within the first 2 to 3 therapy visits, have a diagnosis of shoulder pain, be 18-64 years old, no corticosteroid treatment within the last two weeks, post-surgical cases will be excluded, and patients may not be pregnant. Upon agreeing to the study, patients will sign an informed consent, complete a demographics questionnaire, and complete specific outcome measure assessments. The outcome measures will include the Numeric Pain Rating Scale (NPRS) and the Penn Shoulder Score (PENN). After completing the initial paperwork, patients will be randomized into two groups, control and intervention. The Control group will receive standard FUNHAB® in-office care in addition to standard TB-KT taping technique. The Intervention group will receive standard FUNHAB® in-office care plus varying tension application of TB-KT. The TB-KT will be applied to the shoulder complex to influence proper activation of the rotator cuff muscles, specifically the supraspinatus and infraspinatus. The tape will be applied in an "I" strip from the vertebral border of the scapula to the lesser tubercle of the humerus. Over the course of the 4 weeks, the tension of the tape will systemically increase. At the beginning of each week the tape will be reapplied, and pain rating will be recorded. At the conclusion of 4 weeks patients will complete the PENN.

ELIGIBILITY:
Inclusion Criteria:

* tested within the first 2 to 3 therapy visits, have a diagnosis of shoulder pain, and be 18-64 years old

Exclusion Criteria:

* Corticosteroid treatment within the last two weeks, post-surgical cases, and pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jena Slaski, MEd, ATC, Study Director — Sport and Spine Rehab Clinical Research Foundation
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Increasing Tension: The kinesiology tape will be applied to the shoulder complex to influence proper activation of the rotator cuff muscles, specifically the supraspinatus and infraspinatus. The clinician applied the tape in an "I" strip from the vertebral border of the scapula to the lesser tubercle of the humerus. Over the course of the 4 weeks of care, the tension of the Intervention Group's tape will systemically increase based on the following timelines:
  Week 1: 0% tension Week 2: 25% tension Week 3: 50% tension Week 4: 75% tension
  TheraBand Kinesiology Tape: Kinesiology taping technique is designed to target muscles and lymphatic system. Limited research is available for specific conditions, including low back pain, but it is theorized to correct muscle function by inhibiting or facilitating the muscle, improve blood flow, reduce pain, and improve joint alignment.
Period: Overall Study
Arm/Group | Increasing Tension | Control Tension
Started | 16 | 20
Completed | 13 | 12
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Increasing Tension | Control Tension | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Full Range); unit: years] | 42.38 [18 to 63] | 37.75 [19 to 64] | 39.81 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Rate the pain on a scale of 0 to 10, 0 being none and 10 being the worst imaginable pain
Time Frame: Assessed at baseline, 1,2,3, and 4 weeks
Population: Population analyzed based off of the number of subjects who completed the study, see Overall Study Participant Flow section
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Increasing Tension | Control Tension
Number analyzed (Participants) | 13 | 12
units on a scale
  Baseline Pain (T1) | 5.458 (.764) | 5.115 (.734)
  1 Week Pain (T2) | 4.708 (.732) | 3.808 (.704)
  2 Week Pain (T3) | 3.458 (.663) | 3.115 (.637)
  3 Week Pain (T4) | 3.392 (.641) | 2.923 (.615)
  4 Week Pain (T5) | 2.833 (.588) | 2.269 (.565)

2. Primary Outcome: Penn Shoulder Score (PENN)
Description: The PENN is a outcome measure designed to determine the amount of disability patients are experiencing doing day to day activities. The total score is out of 100, 100 being no disability and 0 being completely disabled.
Time Frame: Assessed at baseline, 1,2,3, and 4 weeks
Population: Population analyzed based off of number of subjects who completed the study, see Overall Study Participant Flow section
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Increasing Tension | Control Tension
Number analyzed (Participants) | 13 | 12
units on a scale
  Baseline PENN (T1) | 53.525 (6.240) | 52.092 (5.995)
  1 Week PENN (T2) | 60.283 (5.220) | 62.646 (5.015)
  2 Week PENN (T3) | 61.742 (5.629) | 67.362 (5.408)
  3 Week PENN (T4) | 65.642 (4.721) | 73.231 (4.536)
  4 Week PENN (T5) | 69.100 (4.958) | 75.873 (4.763)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Increasing Tension | Control Tension
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 0/16 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes